CLINICAL TRIAL: NCT05012852
Title: A Two-part Study; Consisting of a Pilot Part Followed by a Randomized, Parallel Group Part; Comparing Topically Applied Novel Gel Containing Lactic Acid With no Treatment on Women With Candida Vulvovaginitis
Brief Title: Evaluation of VagiVitalAC for Treatment of Candida Vulvovaginitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PepTonic Medical AB (Industry)
Collaborators: StatCons (Unknown); Karolinska Trial Alliance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VagiPep102; CIV-21-06-037087 (Registry Identifier: EUDAMED)
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Vaginal Candidiasis; Vulvovaginal Candidiasis; Candidal Vulvovaginitis
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Intervention Model Description: An single group pilot sub-study followed by a randomized, parallel, controlled sub-study. In the randomized part, the non cured patients in the control goup are given an option to change to active treatment after 7 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VagiVitalAC (Experimental)
  Interventions: Device: VagiVitalAC
- No treatment (No Intervention)

INTERVENTIONS:
Device: VagiVitalAC — In the Pilot part, the single intervention used is VagiVitalAC treatment for 30 days. In the randomized part, patients in the Interventional arm are treated with VagiVital AC for up to 90 days.
  Arms: VagiVitalAC

SUMMARY:
Candidiasis is an infection caused by a yeast (a type of fungus) called Candida. Candidiasis in the vagina is commonly called a "vaginal yeast infection." Another names for this infection is "vaginal candidiasis". The symptoms of vaginal candidiasis include: Vaginal itching or soreness, Pain during sexual intercourse, Pain or discomfort when urinating and Abnormal vaginal discharge. VagiVitalAC is a modified version of the existing gel VagiVital, formulated to act as a treatment for fungal infections.

This clinical investigation is a two-part study consisting of a pilot part followed by a randomized part. The aim of the pilot part is to evaluate if VagiVitalAC is able to cure the vulvovaginal candidiasis in at least 70% of the patients after 7 days treatment. If the proportion of cured patients is at least 70 %, the next part, the randomized part, will be performed. In the randomized part, the treatment efficacy and safety of VagiVitalAC on candida vulvovaginitis will be evaluated by comparing a treatment group with a control group receiving no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be a female, 18 years or older.
* Signed informed consent form.
* Women with earlier recurrent verified vaginal candidiasis.
* Has seeked treatment for suspected fungal infection.
* Be judged by an investigator as having an ongoing vulvovaginal candidiasis.
* If of child-bearing potential, willing to use a reliable method of contraception during the duration of the study. The following methods of contraception are considered reliable: an intrauterine device or any of the following hormonal contraceptives: contraceptive pills, implants, transdermal patches, vaginal ring, injections with prolonged release. A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Be in general good health, as judged by an investigator.

Exclusion Criteria:

* Be currently hospitalized.
* First time with a vulvovaginal candidiasis infection.
* Have a history of ongoing cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, or musculoskeletal disease or disorder that is clinically significant in the opinion of the Principal Investigator or Sub-Investigator.
* Have a history of undiagnosed vaginal bleeding.
* Have an ongoing urogenital infection at the screening visit, other than vulvovaginal candidiasis.
* Any contraindication to the gel (VagiVitalAC) therapy and allergy to the use of any components of the investigational device.
* Pregnant, as determined by urine pregnancy test.
* Have been giving birth during the last 30 days.
* Have a history of drug and/or alcohol abuse within one year of start of study.
* Patient who are currently menstruating or anticipate they will start menstruating within 7 days of starting using the investigational device.
* Have used any intravaginal or systemic antifungal medication within the previous 7 days or had used any intravaginal product such as a spermicide, medicated douche or feminine spray within two days before the start of the study.
* Current treatment for any medical condition that include systemic antimycotics or immunosuppressive drugs.
* Have any reason, which in the opinion of the Principal Investigator would prevent the patient from safely participating in the study or complying with protocol requirements.
* Have participated in another clinical trial within 30 days prior to screening, have received an investigational drug within one month prior to the initial dose of the investigational medical device, or be likely to participate in another clinical trial or receive another investigational medication during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Presence or not of candida fungi in the vaginal culture after 7 days treatment | Day 7

SECONDARY OUTCOMES:
Presence or not of candida fungi in the vaginal culture after 30 days treatment | Day 30
For patients with initial treatment effect (i.e., no presence of candida fungi in the vaginal culture) after 7 days treatment, relapse at day 30, after continued treatment | Day 30
Change in self-reported vulvovaginal symptoms (vaginal itching/burning and/or soreness and/or vaginal discharge and/or pain during sexual intercourse) after 7 days treatment compared to baseline (patient's own experience) | Day 7
Change in self-reported vulvovaginal symptoms after 7 days treatment compared with baseline (patient's own experience), that has been self-identified by the patient as being the most bothersome to her | Day 7
Change in self-reported vulvovaginal symptoms (vaginal itching/burning and/or soreness and/or vaginal discharge and/or pain during sexual intercourse) after 30 days treatment compared to baseline (patient's own experience) | Day 30
Change in self-reported vulvovaginal symptoms after 30 days treatment (patient's own experience), that has been self-identified by the patient at baseline as being the most bothersome to her | Day 30
Frequency of Adverse events Adverse Events (AEs)/Serious Adverse Events (SAEs)/Device Deficiencies (DDs)/Adverse Device Effects (ADEs)/Serious Adverse Device Effects (SADEs) at 7 days | Day 7
Frequency of Adverse events AEs/SAEs/DDs/ADEs/SADEs at 30 days | Day 30
Presence or not of candida fungi in the vaginal culture after 90 days treatment. | Day 90
  Only applicable for randomized part
For patients with initial treatment effect by VagiVitalAC (i.e. no presence of candida fungi in the vaginal culture) after 7 and 30 days treatment, relapse at day 90, after continued treatment. | Day 90
  Only applicable for randomized part
Change in self-reported vulvovaginal symptoms after 7 days treatment compared to baseline, Investigational device group compared to comparator group (patient's own experience). | Day 7
  Only applicable for randomized part
Change in self-reported vulvovaginal symptoms after 7 days treatment, Investigational device group compared to comparator group (patient's own experience), that has been self-identified by the patient at baseline as being the most bothersome to her. | Day 7
  Only applicable for randomized part
Change in self-reported vulvovaginal symptoms (vaginal itching/burning and/or soreness and/or vaginal discharge and/or pain during sexual intercourse) after 90 days treatment compared to baseline (patient's own experience). | Day 90
  Only applicable for randomized part
Change in self-reported vulvovaginal symptoms after 90 days treatment (patient's own experience), that has been self-identified by the patient at baseline as being the most bothersome to her. | Day 90
  Only applicable for randomized part
Frequency of Adverse events AEs/SAEs/DDs/ADEs/SADEs at 7 days, Investigational device group compared to comparator group | Day 7
  Only applicable for randomized part
Frequency of Adverse events AEs/SAEs/DDs/ADEs/SADEs at 90 days. | Day 90
  Only applicable for randomized part

CONTACTS AND LOCATIONS:
Overall Officials: Aino Fianu Jonasson, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No